CLINICAL TRIAL: NCT06162806
Title: Evaluation of Adding Magnesium Sulfate to (Fentanyl/Bupivacaine)Bi-mixture as an Adjuvant to Local Anesthesia in Caudal Block Among Pediatrics in Lower Abdominal Urological Surgeries. a Prospective Randomized Comparative Study
Brief Title: Evaluation of Adding Magnesium Sulfate to (Fentanyl/Bupivacaine)Bi-mixture in Caudal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abd elmoneim Adel Abd elmoneim, clinical professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS-454-2022
Record Dates: First submitted 2023-09-23; First posted 2023-12-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): This group of patients will receive ultrasound guided caudal epidural block using 1ml/kg of Bupivacaine +0.5ulkg fentanyl
  Interventions: Procedure: ultrasound guided caudal epidural block using 1ml/kg of Bupivacaine 0.25% + 0.5microgram/kg of Fentanyl
- Group B (Experimental): This group of patients will receive ultrasound guided caudal epidural block with 50 mg of magnesium added to (1ml/kg Bupivacaine+0.5ulkg fentanyl)bi-mixture
  Interventions: Procedure: ultrasound guided caudal epidural block using 50 mg of Magnesium sulfate added to(1ml/kg of Bupivacaine 0.25% + 0.5microgram/kg of Fentanyl)

INTERVENTIONS:
Procedure: ultrasound guided caudal epidural block using 1ml/kg of Bupivacaine 0.25% + 0.5microgram/kg of Fentanyl — injection of local anesthetic mixture(Bupivacaine +Fentanyl ) in the caudal epidural space under guidance of ultrasound, it is performed by inserting a needle through the sacral hiatus to gain entrance into the sacral epidural space
  Arms: Group A
Procedure: ultrasound guided caudal epidural block using 50 mg of Magnesium sulfate added to(1ml/kg of Bupivacaine 0.25% + 0.5microgram/kg of Fentanyl) — injection of local anesthetic mixture(Bupivacaine +Fentanyl +magnesium sulfate) in the caudal epidural space under guidance of ultrasound, it is performed by inserting a needle through the sacral hiatus to gain entrance into the sacral epidural space
  Arms: Group B

SUMMARY:
this is a randomized controlled study ,patients will be randomly divided into 2 groups , Group A will receive caudal block using 1ml/kg Bupivacaine +0.5u/kg fentanyl, Group B will receive caudal block 50 mg magnesium sulfate added to (1ml/kg Bupivacaine +0.5u/kg fentanyl)

DETAILED DESCRIPTION:
A total of 50 pediatric patients undergoing lower abdominal urological surgeries will be enrolled in this prospective randomized controlled (RCT) study.

I- Randomization:

All included subjects will be randomly allocated and will be divided into two groups; (Group A): will receive [Fentanyl / Bupivacaine], and (Group B): will receive magnesium sulfate added to the previous bi-mixture [Fentanyl / Bupivacaine]. Using computer generated number and concealed using sequentially numbered, sealed opaque envelope technique. There will be no restrictions or stratiﬁcation in the randomization process. The allocation envelope will be opened by the assistant lecturer at the time of anesthetic preparation. Also, the drug preparation will be conducted by an anesthetist who will not involve in any of the study collection data. Finally, the data will be analyzed on an intention-to-treat basis and included all patients who were randomly assigned.

II- Study protocol

1. Pre-operative preparation All children will be anaesthetized in accordance with the local policy of the Abou El-Resh pediatric hospital-Cairo University's pediatric anesthetic unit. Except for oral clear fluid intake 2 hours before surgery, all children will fast for 6 hours. Patients will attend in the preparation room one hour before the operation to get a preoperative checkup, their age and body weight will be recorded as well.
2. Intra-operative management

Premedication by intramuscular injection of atropine 0.02 mg/Kg and midazolam 0.2 mg/Kg will be followed by insertion of intravenous (I.V) cannula.

General anesthesia will be induced in supine position under standard basic monitoring of vital signs with inhalational anesthetic using (100%) O2 + Sevoflurane. After deepening of the anesthesia, atracurium 0.5mg/kg and fentanyl 1μg/kg patients will be given, Endotracheal intubation will then follow by appropriate size of endotracheal tube. volume control ventilation (VCV) 5-7 ml/kg and respiratory rate will be adjusted to keep and PaCO2 levels between 30-35 mmHg using (G.E-Datex-Ohmeda, Avance CS2, USA) anesthesia machine. Anesthesia will be maintained with isoflurane 1 MAC with 50% oxygen in air, and atracurium top-ups of 0.1mg/kg will be given every 30 minutes for neuromuscular blockade.

Technique

After induction of anesthesia, each child will be placed in the left decubitus position with hips flexed at 90 degrees, under complete aseptic precautions, disinfecting the back with chlorhexidine and alcohol, then identification of sacral hiatus is attempted by palpation.

By the aid of US, using a linear transducer placed transversely at the midline to obtain the transverse view of sacral hiatus. Between the sacral cornua are two band-like hyperechoic structures; the superficial one is the SCL, and the deep one is the dorsal surface of sacral bone. The sacral hiatus is the hypoechoic region between the 2 band-like hyperechoic structures. At this level, the ultrasound transducer is rotated 90 degrees to obtain the longitudinal view of sacral hiatus.

Under longitudinal view, the block needle is inserted using the "in-plane" technique. it is suggested that advancement of needle tip beyond the apex of sacral hiatus be limited to 5 mm to avoid dural puncture because the distance between the apex of sacral hiatus and dural sac termination can be as short as less than 6 mm. [8]

(Group A):

Patients in this anesthetic group will receive 0.5 µ/kg fentanyl + 1ml/kg Bupivacaine 0.25% (Group B): Patients in this anesthetic group will receive 50 mg magnesium added to the (0.5 µ/kg fentanyl +1ml/kg Bupivacaine 0.25%) Bi-mixture.

After receiving caudal block the patient will be turned to the supine position and surgical incision will be allowed to be done after 15 minutes.

Continuous recording of heart rate, blood pressure, oxygen saturation and respiratory rate will be carried out from the moment of injection at timely intervals intraoperative. Pain assessment using FLACC score will then follow till 12 hours post-operative.

The time passed between the entrance of the needle into the skin and the injection's completion is referred to as caudal block performance time.

If there is an increase in heart rate or mean arterial pressure of 20% of the baseline values after skin incision, then it will be considered as a failed block and these patients will be excluded from the study and fentanyl of 1µ/kg will be given to provide analgesia

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients aging from 2-12 years
* undergoing lower abdominal urological surgeries not exceeding 3 hours
* ASA I and II

Exclusion Criteria:

* parents refusal to participate in the study
* deformities in the spine
* coagulopathy
* localized infection at site of needle insertion
* known allergic to any of the used drugs

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
time to first requirement of rescue analgesia | 24 hours
  the time after the operation when the patient need rescue analgesia

SECONDARY OUTCOMES:
postoperative opioid analgesia consumption | 24 hours
  the total amount of opioids consumed by the patient postoperative
complications | 24 hours
  occurrence of any postoperative complications related to the caudal block

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H Farouk, lecturer, Study Director — Anesthesia department , cairo university; sherif M soaida, assprofessor, Principal Investigator — Anesthesia department , Cairo university
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No